CLINICAL TRIAL: NCT03637452
Title: Baby Albert: Electronic Cigarette Pharmacokinetics (PK) and Abuse Liability
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 8988
Record Dates: First submitted 2018-06-28; First posted 2018-08-20 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Tobacco Use
Keywords: e-cigarettes; juul brand e-cigarette; njoy brand e-cigarette; evolv/mirage DNA 75c brand e-cigarette
MeSH Terms: conditions — Tobacco Use; Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — During their PK (Pharmacokinetics) visits, Blood will be collected during specific time points and plasma will be extracted from the blood. Plasma will be used to analyze the levels of nicotine in it.
  Urine will be collected from female participants in order to confirm their pregnancy status. Saliva will be collected during their screening visit to analyze for cotinine levels in order to check their smoking status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exclusive cigarette smokers: Exclusive cigarette smokers must smoke at least 10 cigarettes per day for the past three months and have exhaled carbon monoxide (eCO) levels of at least 6 ppm at the screening visit.
- Dual (Electronic cigarette and cigarette smoking) users: Dual e-cigarette and cigarette users must have smoked at least 5 cigarettes per day for the last 3 months and use e-cigarettes at least 15 days per month for the last 3 months.

SUMMARY:
The overall aim of the current research is to understand purchasing and product choice behaviors of tobacco/nicotine users if banning the sale of fully nicotinized cigarettes were to go into effect. A sample of up to 30 current cigarette users (n=15) and dual e-cigarette and combustible cigarette users (n=15) who are willing to try an alternative nicotine-delivery device will be recruited. They will complete the screening visit, visit 1 and 2 preceded by 12 hours of nicotine/tobacco abstinent.

DETAILED DESCRIPTION:
Participants will be provided information about the study and will provide initial consent for screening via an online screener. Written consent will be completed in person when participants are present to the laboratory. Eligible participants will include anyone over the age of 18 years and those who exclusively use combustible cigarettes or those who dual use e-cigarettes and combustible cigarettes. For the exclusive cigarette group, we will allow some e-cigarette experimentation. Participants will complete three in-lab study visits (1 screener visit and 2 study visits) separated by a standard minimum 48-hour washout period. They will be offered an Uber or other rideshare service as transportation to each study visit, however, they will not be required to use the service.

Participants will complete an in-person screening visit in which they will be rescreened according to the eligibility criteria. Their exhaled carbon monoxide (eCO) will be checked prior to their visits as well as breath alcohol and urine pregnancy (for females) test will be conducted. Participant will also complete baseline assessment measures and Balloon Analog Risk Task (BART)- computerized task measuring impulsivity. At visit 2, participants will complete a standard 10 puff bout with the three e-cigarette devices and their usual brand cigarette. During visit 3, participants will complete three concurrent choice tasks in a counter-balanced fashion.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years old
* live within 30 miles of the research site
* interested in/willing to use an e-cigarette during study visits
* be willing and able to complete study procedures including specimen collection, survey completion, and remaining nicotine abstinent for 12 hours prior to each study visit
* speak and understand English
* willing to provide informed consent
* bring usual brand cigarettes to screener study visit
* should have healthy veins

Additional Inclusion criteria for smokers:

* smoke at least 10 cigarettes per day for the past three months
* exhaled more than equal to 6 ppm carbon monoxide at the screener visit

Additional Inclusion criteria for dual users:

* smoke more than equal to 5 tobacco cigarettes per day for the last 3 months
* use e-cigarettes at least 15 days per month for the last 3 months, and
* bring e-cigarette device to screener study visit

Exclusion Criteria:

* currently suffering from lung disease including asthma, cystic fibrosis (CF), or chronic obstructive pulmonary disease (COPD), unless it is well-controlled
* currently pregnant or breast-feeding or have plans to become pregnant or begin breast-feeding at any point during the study
* intoxicated at study visits (breath alcohol testing and clean urine drug screen)
* any known allergies or sensitivity to the known major constituents contained in the aerosol of the study e-cigarette devices (e.g., flavorants, vegetable glycerin, propylene glycol)
* User of zero-nicotine e-cigarettes
* history of cardiac event or distress within the past 3 months
* currently suffering from any blood disorder that includes von willebrand, hemophilia, anemia, sickle cell, leukopenia, thrombocytopenia
* currently taking an anticoagulant or blood thinning medications
* have stent, graph, mastectomy or artificial hardware placed in arms or hands (bilaterally)

Additional Exclusion criteria for smokers:

* have previously used any e-cigarette device (cig-a-like, pen style, mod, APV) for longer than 30 days
* use of an e-cigarette device over the past 14 days.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A sample of up to 30 current cigarette smokers and dual e-cigarette and cigarette users who are willing to use/try an alternative nicotine-delivery device will be recruited via advertisements/ recruitment materials (e.g., craigslist, ads on OSU, OU, and UCO campuses, OUHSC, email) and referrals. Participants will live in the Oklahoma City, OK metro area. Participants will be provided information about the study and provide initial consent for screening via an online screener.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Nicotine delivery measured by serum (blood) nicotine | 1 month
  Participants will complete one standardized puffing bout (10 puffs) with each of the three electronic cigarettes and their usual brand cigarette. Serum nicotine will be measured throughout each standardized puffing bout. Greater levels of serum nicotine will be indicative of greater nicotine delivery.
Proportion of puffs earned and allocated to each product in three hypothetical tobacco regulatory scenarios | 1 month
  Participants will complete three computer tasks simulating hypothetical regulatory scenarios and will earn and allocate puffs to study products. A greater proportion of puffs allocated will indicate greater demand for the product in that hypothetical scenario

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Wagener, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center Tobacco Research Center, Oklahoma City, Oklahoma, United States